CLINICAL TRIAL: NCT06566807
Title: Oxygen Study-Orelabrutinib Combined With Obinutuzumab(O2) for First-Line Treatment of Marginal Zone Lymphoma: A Phase 2, Single-Arm, Prospective, Multicenter Clinical Study
Brief Title: Oxygen Study-Orelabrutinib Combined With Obinutuzumab(O2) for First-Line Treatment of Marginal Zone Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huai'an First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2024-180-01
Record Dates: First submitted 2024-08-14; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Marginal Zone Lymphoma
Keywords: orelabrutinib; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — orelabrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- O2 (Experimental)
  Interventions: Drug: Orelabrutinib, obinutuzumab

INTERVENTIONS:
Drug: Orelabrutinib, obinutuzumab — orelabrutinib，150mg，D1-D28 obinutuzumab，1000mg，D1、D8、D15/cycle1 D1/cycle2-6 . The patients will be treated with 6 cycles of O2 regimen. Patients with CR/PR after 6 cycles of O2 treatment will be treated with 1 year of single-agent orelabrutinib regimen.

SUMMARY:
This is a multi-center, prospective study. The main purpose is to evaluate the efficacy and safety of Orelabrutinib combined with Obinutuzumab for previously untreated MZL.

DETAILED DESCRIPTION:
Marginal zone lymphoma (MZL) is a relatively common type of B-cell non-Hodgkin lymphoma (B-NHL), with an incidence rate second only to diffuse large B-cell lymphoma (DLBCL) and follicular lymphoma (FL). It is divided into three subtypes based on different clinical manifestations and pathological characteristics: mucosa-associated lymphoid tissue lymphoma (MALT), also known as extranodal marginal zone lymphoma, nodal marginal zone lymphoma (NMZL), and splenic marginal zone lymphoma (SMZL). Currently, there is no unified and standardized treatment plan for newly diagnosed MZL. Although high-intensity immunochemotherapy regimens have a high remission rate, they also bring higher treatment-related safety risks. Therefore, exploring effective chemotherapy-free regimens for MZL patients is an attempt with scientific value and clinical significance. With the development of new drugs, new drug regimens have become prominent in the treatment of MZL, and there is an increasing amount of research data on BTK inhibitors in the field of MZL. The BTK inhibitor Orelabrutinib has shown good efficacy in MZL and has been approved by the NMPA for the treatment of MZL in patients who have received at least one prior treatment.

This study is a multi-center, prospectivet clinical study for previously untreated MZL.

The patients will be treated with 6 cycles of O2 regimen. Patients with CR/PR after 6 cycles of O2 treatment will be treated with 1 year of single-agent orelabrutinib regimen.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years, gender not limited;
* Histopathologically confirmed CD20-positive marginal zone lymphoma including MALT, SMZL, NMZL;
* MZL that has progressed, recurred, or is not suitable for local treatment after previous local treatment (local treatments include surgery, radiotherapy, Helicobacter pylori treatment, and hepatitis C treatment);
* ECOG 0-2;
* Indication for treatment as judged by the investigator (symptomatic, with cytopenia, at risk of end-organ damage, bulky disease, persistent progression, or patient's desire for treatment);
* Major organ function meets the following criteria: a) Complete blood count: Absolute neutrophil count ≥1.5×10^9/L, platelets ≥75×10^9/L, hemoglobin ≥75g/L; if accompanied by bone marrow invasion, absolute neutrophil count ≥1.0×10^9/L, platelets ≥50×10^9/L, hemoglobin ≥50g/L; b) Blood biochemistry: Total bilirubin ≤1.5 ULN, AST or ALT ≤2 ULN; serum creatinine ≤1.5 ULN; serum amylase ≤ULN; c) Coagulation function: International normalized ratio (INR) ≤1.5 ULN.
* Expected survival time ≥3 months;
* Voluntarily sign a written informed consent form before the trial screening.

Exclusion Criteria:

* Currently or previously diagnosed with other malignant tumors, unless curative treatment has been performed and there is evidence of no recurrence or metastasis within the last 5 years;
* Lymphoma involving the central nervous system or transformation to a higher grade;
* Active bleeding within 2 months prior to screening, or currently taking anticoagulant medications, or the investigator considers there to be a definite bleeding tendency;
* Major surgery within 6 weeks prior to screening or minor surgery within 2 weeks prior to screening;
* Active infection or uncontrolled HBV (positive for HBsAg and/or HBcAb and positive for HBV DNA titer), HCV Ab positive, HIV/AIDS, or other serious infectious diseases;
* Any mental or cognitive disorder that may limit the understanding, execution, and compliance with the informed consent form and the study;
* Pregnant or lactating women and women of childbearing age who are unwilling to take contraceptive measures;
* Need to continuously take drugs with moderate to severe inhibitory or strong inductive effects on cytochrome P450 CYP3A;
* Other conditions that the investigator considers unsuitable for participating in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2026-08-10 (Estimated); Study Completion 2028-08-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | At the end of Cycle 6 (each cycle is 28 days)
  The ORR is defined as the proportion of patients with a response of CR or PR

SECONDARY OUTCOMES:
the complete response rate | (up to 2 year)
  CRR is defined as the proportion of patients with a response of CR
BOR | Up to 2 years
  The BOR is defined as the proportion of patients with a best response of CR or PR
Duration of Response (DOR) | [ Time Frame: Up to 3 years ]
  Duration of response as defined as the period from the first response (at least PR) to treatment until evidence of disease progression, relapse or death of any cause.
TTR | [ Time Frame: Up to 3 years ]
  TTR is defined as the time from registration to the first response.
24-month time to CR TTCR24 | Up to 2 years
  TTCR24 is defined as the time from registration to the first complete response Within 24 months.
CR at 24 months (CR24) | at 24 months
  CR24 is defined as the proportion of patients with a response of CR at 24 months
2 years progression-free survival | [Time Frame: From date of signing the informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years]
  Progression free survival (PFS) is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment.
2 years overall survival | [Time Frame: From date of signing the informed consent until the date of death from any cause, whichever came first, assessed up to 2 years]
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
The occurrence of adverse events | One month after discontinuation of treatment
  Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University#Huai'an First People's Hospital#, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No